| 1 | The effects of subanaesthetic S-ketamine on postoperative delirium and |
|---|---|
| 2 | cognitive function in elderly patients undergoing non-cardiac thoracic |
| 3 | surgery: a protocol for a randomised, double-blinded, placebo- and |
| 4 | positive-controlled, non-inferiority trial |
| 5 | (SKED Trial) |
| 6<br>7 | |
| 8 | Identifier: NCT05242692 |
| 9 | |
| 10 | |
| 11 | Data of the decomposity loss 4, 2022 |
| 12 | Date of the document: June 1, 2022 |
| 13 | |
| 14 | |
| 11 | |
| 15 | |
| 1.0 | |
| 16 | |
| 17 | |
| 18 | |
| 19 | |
| 13 | |
| 20 | |
| 0.1 | |
| 21 | |
| 22 | |
| 23 | |
| 24 | |
| Δ I | |
| 25 | |
| 0.0 | |
| 26 | |

- 1 The effects of subanaesthetic S-ketamine on postoperative delirium and
- 2 cognitive function in elderly patients undergoing non-cardiac thoracic
- 3 surgery: a protocol for a randomised, double-blinded, placebo- and
- 4 positive-controlled, non-inferiority trial
- 5 (SKED Trial)
- 6 Introduction
- 7 Postoperative delirium (POD) is a neuropsychiatric disorder in elderly
- 8 patients, manifested as an acute onset of altered and fluctuating
- 9 consciousness, inattention, and disorganised thinking. POD occurs in hospital
- up to 1 week postoperatively or until discharge (whichever occurs first), and
- typically the highest incidence is observed during the first 72 hours. [1] The
- incidence of POD varies between 4% to 60%, depending on the age and
- surgical type, although its incidence is underestimated since the hypoactive
- subtype is not well appreciated. [2-7] Postoperative delirium is associated with
- prolonged hospital stay, long-term cognitive and social dysfunction, and even
- death. [8-10] The 1-year survival probability is reduced by approximately 10%
- for each additional day of postoperative delirium. [11] The pathophysiological
- mechanisms of delirium have not been well-elucidated, and
- 19 neuroinflammation remains a topic of mainstream research interest.
- Furthermore, its development results from the complicated interaction of
- 21 multifactorial risks, such as pain, opioids, sleep deprivation, and inflammation,
- which poses a challenge for the prevention and treatment of postoperative
- delirium. [12] Although various techniques, including multi-component non-
- pharmacological interventions, are suggested to reduce the risks, there is
- limited pharmacological methods to reduce the incidence of delirium. [13]
- Dexmedetomidine is a highly selective  $\alpha$ -2 adrenergic receptor agonist that
- is associated with sedative, sympatholytic, and anti-inflammatory effects, and
- has the highest-ranking possibility of preventing postoperative delirium in a

- recent network meta-analysis. [10] Furthermore, the plausibility of
- 2 dexmedetomidine's positive effects on postoperative delirium is enhanced by
- 3 evidence of less anticholinergic activity and opioid-sparing properties. [14]
- 4 Postoperative prophylactic low-dose dexmedetomidine could remarkably
- 5 reduce the incidence of delirium during seven days after non-cardiac surgery;
- 6 [15] moreover, perioperative infusion of dexmedetomidine halved the
- 7 incidence of delirium in the elderly after major cardiac and non-cardiac
- 8 surgery without the increase in adverse effects. [16,17] A randomised
- 9 controlled trial found that intraoperative dexmedetomidine did not decrease
- postoperative delirium or affect cognitive function in the elderly undergoing
- major non-cardiac surgery. [18] A meta-analysis including 11 RCTs revealed
- that perioperative dexmedetomidine reduced the incidence of POD in elderly
- patients after non-cardiac surgery, but this came at the cost of an increased
- incidence of hypotension and bradycardia. [19] A meta-analysis of 1301
- patients undergoing cardiac surgery revealed that dexmedetomidine
- decreased postoperative delirium. [20] Nevertheless, this meta-analysis
- should be interpreted with caution, because several of the included studies
- did not consider delirium as the primary outcome, the methodology of delirium
- 19 assessment varied, and dexmedetomidine administration was also
- inconsistent, with differing doses and durations. Furthermore, the finding that
- dexmedetomidine prevents postoperative delirium is also controversial. In the
- 22 DECADE trial, continuous infusions of dexmedetomidine, started at induction
- 23 and maintained for 24 hours, failed to reduce delirium in patients recovering
- from cardiac surgery. Notably, dexmedetomidine non-significantly aggravated
- delirium, probably mediated by hypotension. [21] However, the plausibility that
- dexmedetomidine prevents POD should be discussed separately, because
- 27 physiopathology and incidence of delirium is quite different between non-
- 28 cardiac surgery and cardiac surgery (frequent cerebral embolism). The
- 29 heterogenous ways that dexmedetomidine is administrated (pre- or post-
- operative or both, bolus, continuous et al) also complicated the analysis even

1 more. As with all pharmacological treatment options, the side effects of 2 dexmedetomidine are bradycardia and hypotension in a dose-dependent 3 manner, and more strikingly in the elderly; hence, close haemodynamic 4 monitoring is warranted. 5 Ketamine, a non-competitive N-methyl-D-aspartate (NMDA) receptor 6 antagonist, is pharmacologically rationalised as an effective medication for 7 reducing postoperative delirium, probably due to its neuroprotective 8 properties. Under surgical conditions, the enhanced AMPA/NMDA signalling 9 caused by the activation of cytokine receptors, and high mobility group box 1 10 facilitate an increased influx of glutamate in hippocampal neurones, which 11 ultimately promotes glutamate toxicity. [22] Ketamine can mitigate neuronal 12 apoptosis by inhibiting the activation of NMDA receptors and the transduction of excitatory signals. [23] The assumption of ketamine's beneficial effects on 13 14 delirium is also strengthened by evidence of its opioid-sparing and 15 antidepressant effects. Depression and delirium, induced by similar 16 pathophysiological mechanisms, are thought to overlap. [24,25] A small 17 sample size of a randomised controlled trial indicated that a low-dose single 18 bolus of ketamine at induction significantly attenuated delirium after cardiac 19 surgery. However, the PODCAST study showed that low-dose ketamine failed 20 to decrease postoperative delirium, pain, and opioid consumption, and 21 generated a dose-dependent increase in the occurrence of negative 22 experiences. [26] The PRIDe study offered no possibility for ketamine to 23 prevent postoperative cognitive decline, including delirium. [27] Ketamine

S-ketamine is the S (+) enantiomer of ketamine, which has a higher affinity with aspartate receptor and  $\mu$  opioid receptor. The anaesthetic potency of S-ketamine is two-fold higher than that of racemic ketamine, and it has higher in vivo clearance rate characterized by lower incidence of adverse reactions.

[28] Animal experiments showed that S-ketamine, rather than racemic

remains an off-label treatment for treatment-POD with factors that limit

widespread use including its dissociative effects and abuse potential.

24

25

26

27

28

29

- 1 ketamine, could alleviate the injury of hippocampal neurones exposed to
- 2 glutamate in rodents; a subanaesthetic dose of S-ketamine could remarkably
- 3 mitigate neuroinflammation by inhibiting microglia proliferation and TLR4/NF-
- 4 κB signalling pathway activation, which consequently improved
- 5 neurocognitive function. [29,30] Additionally, S-ketamine could promote the
- 6 plasticity of hippocampal neurones and improve the function of neurones in
- the prefrontal and hippocampal neural circuits. [31] A study on healthy
- 8 volunteers showed that S-ketamine exhibited pro-neuroplastic effects on
- 9 hippocampal structure, which may improve cognitive function after surgery.
- 10 [32] Moreover, a recent study on human metabolome revealed that S-
- ketamine decreases the levels of circulating branched chain amino acids
- which inhibit the synthesis and release of serotonin and noradrenaline in the
- brain. Thus, S-ketamine could, in theory, increase the effects of serotonin and
- 14 noradrenaline in the brain, and contribute to the improvement of depression
- and cognitive impairment. [33] Furthermore, we hypothesize that the
- sympathomimetic and analgesic properties of S-ketamine might partially
- explain its non-inferior property for delirium prevention compared to
- dexmedetomidine. Though S-ketamine has stronger potency and lower
- incidence of adverse reactions, the evidence that it reduces the incidence of
- 20 postoperative delirium is fairly insufficient.
- Since the effects of S-ketamine on postoperative delirium are lack of good
- 22 quality evidences, we designed the current prospective, randomised, double-
- blinded, placebo- and positive-controlled, non-inferiority trial to investigate the
- 24 effect of intraoperative prophylactic S-ketamine on postoperative delirium in
- elderly patients undergoing thoracic surgery compared to dexmedetomidine.

#### 26 Methods

27

### Study setting and design

- This study will be conducted at the Cancer Hospital and Institute of
- 29 Guangzhou Medical University (Guangzhou, Guangdong, China, with

- 1 principal investigator [PI] Dr Yonghua Yao). The study activities are expected
- 2 to commence in March 2022 and be completed in December 2023. The study
- design is in accordance with the standard protocol items for randomised trials
- 4 guidelines. The overall schedule is illustrated in Table 1, and the Consolidated
- 5 Standards of Reporting Trials flow diagram is shown in Figure 1. The current
- 6 study protocol is the fifth version.

8 Table 1. Schedule of enrolment, interventions, and assessments for the trial

| | Enrolment | Allocation | Post-allocation | | | Closeout | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Preoperative<br>assessment | Allocation | Before<br>induction | recovery | 4-hour<br>after<br>surgery | 24-hour<br>after<br>surgery | 48-hour<br>after<br>surgery | 72-hour<br>after<br>surgery | 96-hour<br>after<br>surgery | 30-day<br>after<br>surgery | 60-day<br>after<br>surgery |
| TIME POINT | -T₁ | T <sub>0</sub> | T <sub>1</sub> | T <sub>2</sub> | F <sub>1</sub> | F <sub>2</sub> | F <sub>3</sub> | F <sub>4</sub> | F <sub>5</sub> | F <sub>6</sub> | <b>F</b> <sub>7</sub> |
| ENROLMENT: | | | | | | | | | | | |
| Eligibility screen | X | | | | | | | | | | |
| Informed consent | Х | | | | | | | | | | |
| Allocation | | × | | | | | | | | | |
| INTERVENTIONS: | | | | | | | | | | | |
| S-ketamine | | | + | | <b>*</b> | | | | | | |
| Dexmedetomidine | | | + | | <b>*</b> | | | | | | |
| Normal Saline | | | + | | <b>*</b> | | | | | | |
| ASSESSMENTS: | | | | | | | | | | | |
| Postoperative<br>delirium<br>(3D-CAM) | | | | | х | х | х | х | х | | |
| Pain severity<br>(NRS) | | | | | Х | Х | х | | | | |
| Sleep quality<br>(NRS) | | | | | | х | Х | х | х | | |
| Cognitive<br>function<br>(TICS-40) | | | | | | | | | | х | Х |
| Haemodynamic variables | | | <b>—</b> | | | <b>*</b> | | | | | |
| Emergence<br>delirium<br>(RASS) | | | | х | | | | | | | |
| Plasma<br>biomarkers<br>(ACh, BDNF,<br>TNF-α) | | | Х | х | | | | | х | | |

9

## 10 Participant recruitment

### 11 Inclusion criteria

- 12 1. Aged 60 to 90 years old.
- 13 2. Both sexes.

- 1 3. American Society of Anaesthesiologists (ASA) physical status classification I-III.
- 2 4. Diagnosed with pulmonary, oesophageal or mediastinal disorders.
- 3 5. Undergoing open or video-assisted thoracic surgery, including lobectomy,
- 4 segmentectomy, pneumonectomy, oesophagectomy, or resection of the mediastinal
- 5 tumour.
- 6. General anaesthesia with one lung ventilation (OLV) or bronchial blocker.
- 7. An expected operation duration of 2 hours or more.
- 8. Voluntary participation in the trial and signed informed consent.

# 9 Exclusion criteria

- 10 1. History of severe psychiatric disease.
- 11 2. History of glaucoma or hyperthyroidism.
- 12 3. History of severe hepatic (Child-Pugh grade C) or renal (requirement for renal
- 13 replacement therapy) disorders.
- 14 4. Body mass index (BMI) > 35 kg/m<sup>2</sup>.
- 5. Dementia history or baseline Mini-Mental State Examination (MMSE) score of < 23.
- 16 6. Severe audio-visual impairments, or inability to speak Mandarin or Cantonese
- 17 precluding communication.
- 7. Sinus bradycardia (heart rate < 50 beats per minute, bpm), sick sinus or Wolff-
- 19 Parkinson-White syndrome, or 2nd degree atrioventricular block and over.
- 8. Uncontrolled hypertension (baseline value > 200/110 mm Hg).
- 9. Allergic to dexmedetomidine or S-ketamine.
- 22 10. Taking sedatives, antidepressants or glucocorticoids.
- 23 11. Alcohol or Illicit drug misuse disorder.
- 24 12. Life expectancy of less than two months due to extensive tumour metastasis.

#### Participants consent

25

- 27 All patients scheduled for thoracic surgery will be screened one day before
- the operation for eligibility at the preoperative evaluation clinic (or on Friday
- for those who will undergo surgery the following Monday). Eligible patients will

- be informed by the study team coordinator. For the sake of voluntary
- 2 participation, all patients will be informed about the aims, procedures,
- 3 benefits, possible risks of study, and how to react if risks occur. If interested in
- 4 enrolment, the patients or their next of kin will sign the written consent form in

5 triplicate.

6

7

10

12

13

14

15

16

17

18

21

23

25

26

27

28

29

30

#### Randomisation and blindness

8 A randomisation code will be generated in a block size of six on the website of

9 <a href="http://www.Randomization.com">http://www.Randomization.com</a> and kept in a sealed opaque envelope by an

anaesthetist nurse. The patients will be randomly allocated by a ratio of 1:1:1

to the S-ketamine group (S group), dexmedetomidine group (D group), or

control group (C group) by an anaesthetist nurse. Dispensing and labelling of

the study drugs will be performed by a pharmacist. Both the anaesthetist

nurse and the pharmacist will not be involved in the following research or

follow-up. The randomisation protocol will be kept secure by the anaesthetist

nurse. The primary investigator, and the clinicians collecting the data, are

allowed to unmask the randomization protocol only when both recruitment and

the database are closed.

The labelled "Study medication" syringes (50 ml), identical in appearance,

and the infusion regimen formulated by the pharmacist based on the

randomisation, will be distributed to the attending anaesthesiologists

responsible for anaesthetic management as soon as the research team

informs the central pharmacy about the patient heading for surgery. In order

to avoid anaesthesiologists' speculation about the randomised assignment,

the study drugs will be infused at the same rate (see Table 2). The

anaesthesiologists, patients, investigators responsible for follow-up, and

statisticians will be all blinded to the randomised allocations until the final

statistical analyses are completed. The blindness will be unmasked by the

primary investigator in a medical emergency, including deterioration of the

patient's condition intraoperatively or adverse events postoperatively.

2

Standard anaesthetic management

3 On the day of the operation, the patients will be admitted to the operating room after random assignment. Vital signs will be routinely monitored, 4 5 including heart rate (HR), blood pressure (BP), oxyhaemoglobin saturation by 6 pulse oximetry (SpO<sub>2</sub>), end-tidal carbon dioxide partial pressure (EtCO<sub>2</sub>), 7 nasopharyngeal temperature, and urine output throughout surgery. Pre-8 oxygenation with 100% oxygen for 15 min before the induction of anaesthesia 9 will be delivered to the patient using a face mask. Atropine will be 10 administered intravenously in avoidance of excessive secretions. 11 After arterial line and central venous line are cannulated under ultrasound 12 guidance, anaesthesia induction will be performed by administration of 13 midazolam (0.05 mg/kg), propofol (1-2 mg/kg) or etomidate (0.2 mg/kg), and 14 sufentanil (0.2-0.4  $\mu$ g/kg). After the patient becomes unconscious, rocuronium 15 (0.6 mg/kg) will be injected intravenously. Bronchial intubation will be 16 performed smoothly with a video laryngoscope after 3-minute positive 17 pressure ventilation. The tip of double lumen tubes (DLTs) will be inserted into 18 the glottis under direct vision and advanced until a mild resistance is 19 perceived. After the fibreoptic bronchoscope is fully lubricated, it will be 20 advanced into the tracheal lumen of the DLTs until the carina is identified. 21 Afterwards, the ideal position of the bronchial lumen (the blue bronchial cuff 22 should be invisible for left DLTs, the opening in the upper lobe of the right lung 23 should be visible for right DLTs) will be verified. Dual-controlled ventilator 24 modes (i.e. pressure-controlled ventilation with volume guaranteed or 25 pressure-regulated volume control) will be applied. One-lung protective 26 ventilation regimen will be conducted by a combination of tidal volumes (Vt) of 27 6 ml/kg or lower, by predicted body weight, with a positive end-expiratory 28 pressure of 6 cmH<sub>2</sub>O or beyond based upon guidelines and expert opinion for 29 optimal practice during OLV. [34] High inspiratory fractions of oxygen (FiO<sub>2</sub> > 30 70%) will be administered to maintain SpO<sub>2</sub> higher than 94%. In addition,

1 continuous positive airway pressure (CPAP) regimen will be considered when 2 necessary. The respiratory rate will be adjusted to maintain EtCO<sub>2</sub> at 35-45 3 mmHg. Sedative maintenance will be performed with a TCI (target-controlled 4 infusion) of propofol according to the Schnider model at a plasma 5 concentration (Cp) of 2-3  $\mu$ g/ml to maintain the bispectral index value 6 between 40 and 60. Analgesic maintenance will be achieved with a TCI of 7 remifentanil according to the Minto model at a Cp of 1-6 ng/ml to fluctuate the 8 HR and BP within the baseline value ± 20%. An intermittent bolus of 9 rocuronium will be administered to maintain TOF < 1 intraoperatively. Forced 10 air-warm blankets will be used to ensure an intraoperative body temperature 11 of 36-37°C. The surgeon will implement an intercostal nerve block (T3-7) with 20 ml of 0.5% ropivacaine under direct thoracoscopic view before placing a 12 13 chest tube. The sign of a successful block is the presence of pleural 14 displacement. All participants will be given hydromorphone (0.015 mg/kg) 15 when a chest tube is placed for the sake of prophylaxis of hyperalgesia. 16 A patient-controlled analgesia (PCA) device, with hydromorphone (0.15 mg/kg) and ondansetron (12 mg) in a total volume of 100 ml, will be 17 18 connected to the intravenous cannula at the end of surgery. The device is 19 programmed to administer a background dose of 2 ml/h, as well as a bolus 20 dose of 0.5 ml with a lockout interval of 15 min for 48 hours. Hydromorphone 21 (0.008 mg/kg) will be administered if the numeric rating scale (NRS) score is > 22 5 despite the PCA regimen. Residual neuromuscular blockade will be 23 routinely reversed with neostigmine (40  $\mu$ g/kg) and atropine (20  $\mu$ g/kg), and 24 the endotracheal tube will be removed when the patients are able to follow 25 verbal commands. 26 27 Study drugs administration 28 S-ketamine (50 mg, 2 ml) is diluted to 50 ml (1 mg/ml) with 48 ml normal 29 saline; dexmedetomidine (200  $\mu$ g, 2 ml) is diluted to 100 ml (2  $\mu$ g/ml) with 98

ml normal saline; the control group only receives 50 ml normal saline in light

- of blindness. All drugs are identical in appearance, packaged in identical 50
- 2 ml syringes labelled with "Study medications". The loading dose of study
- drugs will be infused within 10 minutes before induction, and the maintenance
- 4 dose will be infused at a constant rate continuously until skin closure. In the
- 5 preliminary trial, we found that a loading dose of 0.4  $\mu$ g/kg
- 6 dexmedetomidine lead to obvious bradycardia and transient hypertension
- 7 events. Therefore, we modified the loading dose of dexmedetomidine to 0.2
- 8  $\mu$ g/kg; In addition, in order to ensure blindness, the infusion speed of
- 9 dexmedetomidine is consistent with that of S-ketamine, which also reduces
- 10 the side effects of dexmedetomidine. The detailed administrative protocol of
- study drugs is shown in Table 2.

13

14

15

16

Table 2 Study drugs and administrative protocol (take a 60 kg patient as an example)

| Group | Concentration | Loading | Maintenance |
|---|---|---|---|
| | | dose | dose |
| S-ketamine | 1 mg/ml | 0.25 mg/kg | 0.1 mg/kg/h |
| i.e. The administrative protocol of a 60 kg patient will be a loading dose | | | a loading dose of |
| 15 ml and a maintenance dose of 6ml/h | | | |
| Dexmedetomidine | 2 <b>µ</b> g/ml | 0.2 <b>μ</b> g/kg | 0.2 <b>µ</b> g/kg/h |
| i.e. The administrative protocol of a 60 kg patient will be a loading dose of | | | |
| 15 ml and a maintenance dose of 6 ml/h | | | |
| Control | Normal saline | | |
| i.e. The administrative protocol of a 60 kg patient will be a loading dose of | | | |
| 15 ml and a maintenance dose of 6 ml/h | | | |

#### Data collection

- 17 The following data will be collected through patient interviews and
- abstractions from the electronic medical record system:

### Preoperative data collection

1

8

- 2 1. Patient demographic data including age (years), sex, height (cm), weight (kg), BMI
- 3 (kg/m²), and education level (years).
- 4 2. ASA classification, Charlson comorbidity index, baseline MMSE, and type of surgery.
- 5 3. Plasma biomarker concentrations including acetylcholine (ACh), brain-derived
- 6 neurotrophic factor (BDNF) and tumour necrosis factor- $\alpha$  (TNF- $\alpha$ ) before the
- 7 administration of study drugs (T1).

## Intraoperative data collection

- 9 1. Haemodynamic parameters including HR (bpm), mean arterial pressure (MAP, mmHg),
- 10 SpO<sub>2</sub> and BIS value at 15-minute intervals.
- 11 2. Hypotension and bradycardia episodes (see Table 3).
- 12 3. Hypertension and tachycardia episodes (see Table 3).
- 13 4. Duration of desaturation (SpO<sub>2</sub> < 94%, minutes).
- 14 5. The cumulative dosage of noradrenaline ( $\mu$ g) and atropine (mg).
- 15  $\,$  6. The consumption of propofol (mg) and opioids (converted to morphine milligram
- equivalent by Global RPH, MME).
- 17 7. Surgery, anaesthesia and OLV duration (minutes).
- 18 8. Time to extubation (minutes, duration from discontinuation of propofol to removal of
- the tracheal tube).
- 20 9. Emergence agitation (Richmond Agitation-Sedation Scale, RASS score  $\geq$  1).
- 21 10. Plasma biomarker concentrations at the end of operation (T2).

### 22 Postoperative data collection

- 1. Incident postoperative delirium between 4 h after surgery and the 4th postoperative day, and
- twice daily from postoperative day 1 to postoperative day 4 (8:00-10:00 am) with an
- interval of at least 6 hours.
- 26 2. Severity and duration of delirium.
- 27 3. Postoperative pain at 4 h, 1 and 2 days after surgery.
- 28 4. Consumption of hydromorphone (mg).
- 29 5. Quality of sleep within 4 days after surgery.
- 30 6. Cognitive function at 30 and 60 days after surgery.

1 7. Plasma biomarker concentrations at the 4<sup>th</sup> day after surgery (T3). 2 Data Safety and Monitoring Committee (DSMB) is consist of three senior 3 anaesthesiologists and one surgeon who are blinded to the study. The DSMB 4 will provide independent oversight of the SKED trial and will review the study 5 data for the participant safety as well as CRF storage. The data will be 6 entered into the Epidata V4.6 database protected by password only 7 accessible to DSMB. Then, the data will be exported from Epidata database 8 to a statistical package for analysis by biostatisticians independent of the 9 study. 10 11 **Outcomes** 12 **Primary outcomes** 13 The primary outcome will be the incidence of postoperative delirium as 14 defined by any positive assessment between 4 h after surgery and the 4th 15 postoperative day. 16 Secondary outcomes 17 The main secondary outcome will be the subtype, severity and duration of 18 postoperative 19 delirium. 20 Other prespecified secondary outcomes will be the incidence of emergence 21 delirium; pain 22 severity at 4 h, 1 and 2 days after surgery; quality of sleep within 4 days after 23 surgery; 24 cognitive function at 30 and 60 days after surgery; plasma biomarker (ACh, 25 BDNF, TNF- $\alpha$ ) 26 concentrations at T1-3; and incidence of adverse events.

Measurement of outcomes

29 Measurement of delirium

27

- 1 Delirium will be assessed using a validated 3-minute diagnostic confusion
- 2 assessment method (3D-CAM Chinese version, with a sensitivity of 84%–99%
- and specificity of 90%–97%) [35,36] or Confusion Assessment Method for the
- 4 Intensive Care Unit (CAM-ICU), for patients who have a tracheal tube or
- 5 underwent tracheostomy. [37] 3D-CAM resolves the four diagnostic features
- of delirium: (1) acute onset and fluctuating course, (2) inattention, (3)
- disorganised thinking, and (4) altered level of consciousness. A patient who
- 8 displays both features 1 and 2, with either feature 3 or 4, will be diagnosed
- 9 with delirium (see Figure 2). [35] Delirium assessments will be performed only
- when patients can be aroused sufficiently with an RASS score of -3 to 4
- (Supplementary Table 1). Patients with postoperative delirium will be
- classified into three subtypes. Hyperactive delirium will be defined when the
- 13 RASS score ranges from 1 to 4; hypoactive delirium will be defined when the
- 14 RASS score ranges from -1 to -3, and mixed delirium will be defined when the
- RASS score ranges from 1 to 4 and -1 to -3 alternatively. The severity of
- postoperative delirium will be rated using the CAM-Severity short-form scale
- 17 (Supplementary Table 2). Mild-to-moderate delirium will be defined as a CAM-
- S score of 3 to 5, while severe delirium will be defined as a CAM-S score of 6
- 19 to 7. **[38]**
- Four investigators who are not involved in perioperative care will be
- responsible for postoperative delirium assessments and will be trained by a
- 22 psychiatrist with regard to symptoms, diagnosis, and treatment of delirium.
- 23 Furthermore, the psychiatrist will explain the protocols of 3D-CAM and CAM-
- 24 ICU in detail, and will perform the simulation training of delirium assessment
- until a kappa value over 0.8 is achieved between investigators and
- psychiatrists. The training process will be repeated every 4-6 months
- throughout the study. In addition, the chart-based delirium identification
- instrument with the information primarily derived from electronic medical
- 29 records system and recalling descriptions of caregivers will be employed to

- detect any cases of delirium in patients that may occur outside of in-person
- 2 delirium assessments (Supplementary Table 3). [39]

# 3 Pain and sleep quality measurement

- 4 Postoperative pain at rest and during a cough will be evaluated using an 11-
- point NRS (0 = [no pain], 0 < NRS < 4 [mild pain],  $4 \le NRS < 7$  [moderate
- pain],  $7 \le NRS < 10$  [severe pain], NRS = 10 [worst pain imaginable]).
- 7 Postoperative sleep quality will also be evaluated using the NRS (0 = best-
- 8 quality sleep, 10 = worst-quality sleep).

## Cognitive function measurement

9

19

27

28

- 10 Postoperative cognitive function will be assessed using the Chinese version of
- the Telephone Interview for Cognitive Status-40 (TICS-40). The TICS-40
- scale used in this study consists of nine items with a maximum score of 40
- points, including the following variables and corresponding points: address (3
- points), current date (5 points), counting backwards (2 points), word-list
- recalling (10 points), subtractions (5 points), object naming (2 points),
- repetition (1 point), the president and prime minister's names (2 points), and
- delayed recall of the word list (10 points). A score below 21 will be defined as
- mild cognitive impairment (Supplementary Table 4). [40]

### Biomarkers concentration measurement

- Venous blood (approximately 6 ml) will be sampled and stored on ice in
- vacutainer tubes containing EDTA. Within 30 min, the samples will be
- 22 centrifuged at 4°C for 20 min at 2000× g to obtain plasma and then stored at -
- 80°C. We will measure ACh, BDNF, and TNF- $\alpha$  levels by enzyme-linked
- immunosorbent assay method (in accordance to manufacturer's instructions).
- The biomarker assay will be performed by a specialist who is blinded to the
- randomization. (Supplementary text for the rationales of biomarkers selected)

### Adverse events

- 29 An adverse event (AE) can be any unfavourable and unintended symptom or
- 30 side effect temporally associated with the use of study medications. The

- 1 potential AEs that may be considered in this trial are bradycardia,
- 2 hypotension, tachycardia, hypertension, arrhythmia, nystagmus,
- 3 hypersalivation, euphoria, emergence agitation, hallucinations, and
- 4 nightmares. It is possible, but very unlikely, that low-dose S-ketamine (50 mg
- 5 in total) administered intraoperatively will cause these psychiatric effects.
- 6 Potential adverse events and medical rescue are shown in Table 3. [41]
- 7 Serious AEs are rare, life-threatening events that may be associated with
- 8 the study drugs or perioperative incidents, such as death or serious cardio-
- 9 cerebral vascular events.

11

# Table 3 The definitions of adverse events and corresponding medication

## 12 rescue

| Adverse events | Severity | Definition | Treatment |
|---|---|---|---|
| Hypotension<br>(SBP<90 mm Hg or<br>DBP<50 mm Hg or<br>MAP<80% baseline) | Mild<br>Moderate<br>Severe<br>Life-<br>threatening | SBP 80-89 mm Hg SBP 70-79 mm Hg>2 min SBP 60-69 mm Hg>1 min SBP 60-69 mm Hg and unresponsive to noradrenaline or SBP<60 mm Hg | Close monitoring Noradrenaline 4 µg \$ Noradrenaline 8 µg # Intensive intervention and suspend the study |
| Hypertension<br>(SBP>140 mm Hg or | Mild | SBP 141-160 mm Hg | Close monitoring |
| DBP>90 mm Hg or<br>MAP>120% baseline) | Moderate | DBP 91-100 mm Hg<br>SBP 160-170 mm Hg | Urapidil 12.5 mg |
| | Severe | or<br>DBP 101-110 mm Hg<br>>3 min<br>SBP 171-180 mm Hg | Urapidil 25 mg or NG 50 $\mu$ g Intensive intervention |
| | Life-<br>threatening | or DBP 111-120 mm Hg >2 min SBP>180 mm Hg or DBP>120 mm Hg and | and suspend the study |

| Bradycardia | Mild | unresponsive to NG<br>HR 55-60 bpm | Close monitoring |
|---|---|---|---|
| (HR<60 bpm) | Moderate<br>Severe | HR 50-54 bpm>3 min<br>HR 40-50 bpm>2 min | Atropine 0.5 mg Atropine 1.0mg |
| | Life- | HR<40 bpm and | Intensive |
| | threatening | unresponsive to | intervention |
| | | atropine | and suspend the study |
| Tachycardia | Mild | HR 90-100 bpm | Close monitoring |
| (HR<60 bpm) | Moderate | HR 101-110 bpm>3 | Esmolol 20 mg |
| | Severe | min | Esmolol 40 mg |
| | Life-<br>threatening | HR 111-130 bpm>2<br>min | Intensive intervention |
| | uncatering | HR>130 bpm and | and suspend the |
| | | unresponsive to | study |
| | | Esmolol | • |
| Hypoxemia | Mild | SpO <sub>2</sub> 90%-94% | Close monitoring |
| (SpO <sub>2</sub> <94%) | Moderate | SpO <sub>2</sub> 80%-90%>3 | CPAP |
| (OPO2 10 170) | Severe<br>Life- | min<br>SpO <sub>2</sub> 70%-79%>2 | Two-lung ventilation |
| | threatening | min | Intensive |
| | unoatomig | SpO <sub>2</sub> <70% and | intervention |
| | | unresponsive to two- | and suspend the |
| | | lung | study |
| | | ventilation | |
| Emergence delirium | Mild | RASS 1-2 | Limb restraint |
| | Severe | RASS 3-4 | Propofol 30 mg |
| Hallucination/Nystagmus | NA | 3D-CAM | Haloperidol 10 mg |

- 3D-CAM, 3 minutes diagnostic confusion assessment method; CPAP,
- 2 constant positive airway pressure; HR, heart rate; NA, not applicable; NG,
- 3 nitro-glycerine; RASS, Richmond Agitation-Sedation Scale.
- \$ followed by continuous infusion with 0.01-0.1  $\mu$ g/kg/min when necessary
- 5 # followed by continuous infusion with 0.1-0.2  $\mu$ g/kg/min when necessary

## Sample size calculation

6

- 8 The sample size was calculated for the main outcome, the incidence of
- 9 postoperative delirium, using PASS software version 11.0. Based on previous
- studies and our recently completed data, we estimated that the incidence of

- 1 POD in elderly patients undergoing non-cardiac thoracic surgery was 40%.
- 2 [12,42-46] Assuming that dexmedetomidine is associated with a 40% relative
- 3 reduction in the incidence of postoperative delirium, the non-inferiority margin
- 4 rate ratio (RR) of S-ketamine versus dexmedetomidine will be set at 1.5.
- 5 [15,27,47,48] To achieve a two-sided type I error of 5% and 80% power, 729
- 6 participants (243 patients per arm) will be recruited. To accommodate a 5%
- dropout rate, the final sample size will be 780 (260 patients per arm).

9

### Statistical methods

- 10 Kolmogorov-Smirnov test will be used to evaluate the normal distribution of
- 11 continuous variables. Normally distributed data will be presented as means ±
- standard deviation (SD), and non-normally distributed data will be presented
- as medians with interquartile ranges. Categorical data will be summarised as
- 14 counts (proportions).
- The absolute standardised difference (ASD) will be used for the comparison
- of baseline data among the three groups, that is, the absolute difference in
- means, mean ranks, or proportions divided by the combined SD. Baseline
- variables with ASD>0.013 (i.e., 1.96  $\times$
- $\sqrt{(260 + 260 + 260)/(260 \times 260 \times 260)}$ ) are considered to be imbalanced
- and will be adjusted for in all analyses when necessary.
- For the primary outcome, the incidence of postoperative delirium, the
- intention-to-treat approach and per-protocol (PP) approach will be performed.
- Pearson's chi-square test will be applied to compare proportions with the
- primary outcome among groups. The difference among groups will be
- expressed as RR and 95% confidence interval (CI), while non-inferiority will
- be identified if the upper limit of 95% CI of RR is < 1.5. For the secondary
- outcomes, only the PP approach will be used. Normally distributed data will
- be analysed with one-way analysis of variance (ANOVA); Non-normally
- distributed data will be analysed with Kruskal-Wallis test. The median

- difference will be calculated using the Hodges-Lehmann estimation on the
- 2 basis of the Kruskal-Wallis test. Adverse events that are presented as
- incidences will be compared by calculating the 95% CI of the incidence
- 4 difference: incidence (S group) incidence (D group), and noninferiority will
- 5 be achieved if the upper limit of 95% CI is < 5%. The superiority for outcomes
- 6 will be assessed when noninferiority is verified.
- 7 To account for correlation among repeated measurements, such as numeric
- 8 rating scores for pain and sleep quality, plasma biomarker concentrations,
- 9 and cognitive function, will be compared using generalised estimating
- equation analysis among groups. The time to delirium will be calculated with
- the Kaplan-Meier estimator, and the differences among groups will be
- 12 assessed by the log-rank test. The number needed to treat will be estimated
- 13 for the primary outcome.
- Missing values will be adjusted using random forest imputation in the
- missForest package. However, missing values, due to fatigue in the
- assessment or the patient's inability to cooperate, will be imputed with positive
- 17 results or means in the corresponding treatment group and time point. If the
- patient did not have a delirium assessment at all (e.g. dropout or death), no
- values will be imputed. The last assessment is used to replace the missing
- value to estimate the incidence of postoperative delirium in patients who are
- discharged or die within 4 days, while the missing value of assessment per
- day does not need to be replaced.
- The P values and CIs reported from one-way ANOVA and Kruskal-Wallis
- test will be considered to illustrate statistical significance if they are less than
- 25 0.017 and 98.3%, respectively, accounting for three pairwise comparisons.
- The family-wise significance and CI levels among the three groups will be set
- at 0.05% and 95%, respectively. For the pain intensity score, a 1.1 decrease
- will be considered the minimal clinically important difference. [49]
- 29 Analyses will be conducted using IBM SPSS version 25.0 (SPSS Software,
- 30 Chicago, IL, USA), R statistics version 4.1.2 (R Project for Statistical

1 Computing), and GraphPad Prism version 8.0 (GraphPad Software, San 2 Diego, CA, USA). 3 **Ethics and confidentiality** 4 5 Ethical approval was obtained from the Institutional Review Board of the 6 Cancer Hospital and the Institute of Guangzhou Medical University 7 (ZN202119). The study has also been registered at Chictr.org.cn with the 8 identifier ChiCTR2100052750. The personal information of the participants 9 will not be disclosed unless authorisation is approved. In addition, each 10 participant will be provided with a unique identity code, the information of 11 which will be properly secured. The CRF and Epidata database will be 12 retained for a minimum of 10 years. 13 14 **Patient and Public Involvement** 15 No patients or public representatives were involved in the design of this trial. 16 17 Dissemination 18 At the end of the trial, we commit to making public disclosure available despite the outcome. Public disclosure will include publication in an appropriate 19 20 journal or oral presentation at an academic meeting. The PI will be considered 21 the first or corresponding author. The investigators who contribute a minimum 22 of four months to the trial will be co-authors; otherwise, they will be 23 acknowledged in the publication. 24 25 **Discussion** 26 Lung cancer ranks first among all malignancies in China, and anatomic 27 pulmonary resection is a major component of multimodal therapy according to 28 the lung cancer guidelines. [12] However, more than 40% of patients 29 undergoing lung cancer surgery are inflicted by severe depression-related 30 psychological suffering postoperatively. [50] Depression is an independent

1 predictor of postoperative delirium in patients who undergo orthopaedic and 2 cancer surgeries. [24] Based on its pharmacological mechanisms and 3 antidepressant effects, we speculate that S-ketamine would be non-inferior to 4 dexmedetomidine in reducing postoperative delirium to some extent in the 5 elderly, with fewer episodes of hypotension or less opioid consumption. 6 Hypotension is pertinent to delirium, and minimisation of intraoperative 7 hypotension episodes is recommended to reduce postoperative delirium. [51] 8 Additionally, the administration of opioids (long-acting opioids in particular) is 9 closely related to postoperative delirium in a dose-dependent manner. Hence, 10 it is critical to abate opioid consumption in order to curtail delirium. [8] 11 Although previous studies have demonstrated that ketamine failed to reduce 12 the incidence of postoperative delirium in patients undergoing major cardiac 13 or non-cardiac surgery, we will deploy a different administrative protocol to 14 evaluate the effect of an isomer of ketamine on postoperative delirium 15 accompanied by dexmedetomidine as a positive comparator and by an 16 optimal sample size. Dexmedetomidine is a highly recommended agent in the 17 prevention and treatment of postoperative delirium; however, it is commonly 18 accompanied by hypotension and bradycardia in the elderly. As the 19 prevention of postoperative delirium is more practical and effective than the 20 treatment itself, creating a means of prevention for delirium is extraordinarily 21 indispensable. We believe that the possible result will be one of the following: 22 (1) S-ketamine will be non-inferior to dexmedetomidine in the prevention of 23 postoperative delirium; meanwhile, more stable haemodynamics, lower 24 postoperative pain severity, or other beneficial secondary outcomes will be 25 observed with S-ketamine intervention. Side effects will be compared between 26 groups, all of which will be our desirables. This suggests that S-ketamine will 27 be an optimal choice for limiting delirium emergence in the elderly, and further 28 studies should be performed to evaluate its effect on long-term cognitive 29 function. (2) S-ketamine will be non-inferior to dexmedetomidine in 30 postoperative delirium prevention with comparable secondary outcomes;

| 1 | however, it will be accompanied by frequent side effects. This indicates that |
|---|---|
| 2 | S-ketamine will be clinically valueless for delirium prevention, which is also |
| 3 | possible in view of the results from previous studies on ketamine (PODCAST |
| 4 | and PRIDe study). (3) S-ketamine will be inferior to dexmedetomidine in the |
| 5 | prevention of postoperative delirium, which is probably because |
| 6 | dexmedetomidine is recognised as the most effective medication for delirium, |
| 7 | and fewer studies have compared the two drugs. |
| 8 | The SKED protocol has many limitations. First, the current trial is launched |
| 9 | at special |
| 10 | time when inclusion may be constrained by local SARS-CoV-2 pandemic. As |
| 11 | such, the |
| 12 | research period may take longer than anticipated. Second, this is a single- |
| 13 | centre study |
| 14 | that exclusively involves thoracic surgery; therefore, the generalisability may |
| 15 | not be |
| 16 | extrapolated. Third, an anticipated non-inferiority margin ratio of 1.5 in our trial |
| 17 | may be |
| 18 | too large, and consequently, the sample size may be underestimated. Fourth, |
| 19 | a dropout |
| 20 | rate of 5% seems a bit low as advert events due to dexmedetomidine may be |
| 21 | higher than |
| 22 | that, if so, we would enlarge the sample size upon approval from the IRB. |
| 23 | |
| 24 | |
| 25 | |

#### References

- 2 1 Evered L, Silbert B, Knopman DS, et al. Recommendations for the nomenclature of
- 3 cognitive change associated with anaesthesia and surgery-2018. Br J Anaesth
- 4 2018;**121**(5):1005-1012.
- 5 2 Schenning KJ, Deiner SG. Postoperative delirium in the geriatric patient. *Anesthesiol.*
- 6 *Clin* 2015;**33**:505–16.
- 7 3 American Geriatrics Society Expert Panel on Postoperative Delirium in Older Adults.
- 8 Postoperative delirium in older adults: best practice statement from the American
- 9 Geriatrics Society. *J Am Coll Surg* 2015;220:136–48.e1.
- 10 4 Rudolph JL, Marcantonio ER. Review articles: postoperative delirium: acute change
- with long-term implications. *Anesth Analg* 2011;**112**:1202–11.
- 12 5 Austin CA, O'Gorman T, Stern E, et al. Association Between
- Postoperative Delirium and Long-term Cognitive Function After Major
- Nonemergent Surgery. *JAMA Surg* 2019;**154(4)**:328-334.
- Wang Y, Lei L, Ji M, Tong J, et al. Predicting postoperative delirium after
- microvascular decompression surgery with machine learning. *J Clin*
- 17 Anesth 2020;**66**:109896.
- 18 7 Migirov A, Chahar P, Maheshwari K. Postoperative delirium and
- neurocognitive disorders. *Curr Opin Crit Care* 2021;**27(6)**:686-693.
- 20 8 Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet
- 21 2014;**383**:911–22.
- 9 Lindroth H, Bratzke L, Purvis S, et al. Systematic review of prediction models for
- delirium in the older adult inpatient. *BMJ Open* 2018;**8**:e019223.
- 24 10 Park SK, Lim T, Cho H, et al. Comparative effectiveness of pharmacological
- interventions to prevent postoperative delirium: a network meta-analysis. Sci Rep
- 26 **2021**;**11**:11922.
- 27 11 Pisani MA, Kong SY, Kasl SV et al. Days of delirium are associated with 1-year
- mortality in an older intensive care unit population. Am J Respir Crit Care Med
- 29 2009;**180**:1092–7.
- 30 12 Wei W, Zheng X, Gu Y, et al. Effect of general anesthesia with thoracic paravertebral

- block on postoperative delirium in elderly patients undergoing thoracoscopic lobectomy:
- a randomized controlled trial. *BMC Anesthesiol* 2022;**22**:1-10.
- 13 Jin Z, Hu J, Ma D. Postoperative delirium: perioperative assessment, risk
- 4 reduction, and management. *Br J Anaesth* 2020;**125(4)**:492-504.
- 5 14 Djaiani G, Silverton N, Fedorko L, et al. Dexmedetomidine versus propofol Sedation
- 6 Reduces Delirium after Cardiac Surgery: A randomized controlled trial. *Anesthesiology*
- 7 2016;**124**:362–68.
- 8 15 Su X, Meng ZT, Wu XH, et al. Dexmedetomidine for prevention of delirium in elderly
- 9 patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial.
- 10 Lancet 2016;**388**:1893–902.
- 11 16 Li CJ, Wang BJ, Mu DL, et al. Randomized clinical trial of intraoperative
- dexmedetomidine to prevent delirium in the elderly undergoing major non-cardiac
- 13 surgery. *Br J Surg* 2020;**107**:e123–32.
- 14 17 van Norden J, Spies CD, Borchers F, et al. The effect of peri-operative
- dexmedetomidine on the incidence of postoperative delirium in cardiac and non-
- 16 cardiac surgical patients: a randomised, double-blind placebo-controlled trial.
- 17 *Anaesthesia* 2021;**76**:1342–51.
- 18 Deiner S, Luo X, Lin HM, et al. Intraoperative infusion of dexmedetomidine for
- prevention of postoperative delirium and cognitive dysfunction in elderly patients
- 20 undergoing major elective noncardiac surgery: A randomized clinical trial. JAMA Surg
- 21 2017;**152**:e171505.
- 22 19 Pan H, Liu C, Ma X, et al. Perioperative dexmedetomidine reduces delirium in elderly
- patients after non-cardiac surgery: a systematic review and meta-analysis of
- randomized-controlled trials. Can J Anaesth 2019;66(12):1489-1500.
- $25\,$   $\,$  20 Duan X, Coburn M, Rossaint R, et al. Efficacy of perioperative dexmedetomidine on
- postoperative delirium: systematic review and meta-analysis with trial sequential
- analysis of randomised controlled trials. *Br J Anaesth* 2018;**121**:384–97.
- 28 21 Turan A, Duncan A, Leung S, et al. Dexmedetomidine for reduction of atrial fibrillation
- and delirium after cardiac surgery (DECADE): a randomised placebo-controlled trial.
- 30 *Lancet* 2020;**396**:177–85.

- 1 22 Safavynia SA, Goldstein PA. The role of neuroinflammation in postoperative cognitive
- dysfunction: moving from hypothesis to treatment. *Front Psychiatry* 2018;**9**:752.
- 3 23 Hudetz JA, Pagel PS. Neuroprotection by ketamine: a review of the experimental and
- 4 clinical evidence. *J Cardiothorac Vasc Anesth* 2010;**24**:131–42.
- 5 24 Elsamadicy AA, Adogwa O, Lydon E, et al. Depression as an independent predictor of
- 6 postoperative delirium in spine deformity patients undergoing elective spine surgery. *J*
- 7 Neurosurg Spine 2017;**27**:209–14.
- 8 25 O'Sullivan R, Inouye SK, Meagher D. Delirium and depression: inter-relationship and
- 9 clinical overlap in elderly people. *Lancet Psychiatry* 2014;**1**:303–11.
- 10 26 Avidan MS, Maybrier HR, Abdallah AB, et al. Intraoperative ketamine for prevention of
- 11 postoperative delirium or pain after major surgery in older adults: an international,
- multicentre, double-blind, randomised clinical trial [published correction appears in
- 13 *Lancet* 2017;**390**:267–75.
- 14 27 Hollinger A, Rüst CA, Riegger H, et al. Ketamine vs. haloperidol for prevention of
- cognitive dysfunction and postoperative delirium: A phase IV multicentre randomised
- placebo-controlled double-blind clinical trial. *J Clin Anesth* 2021;**68**:110099.
- 28 Krystal JH, Charney DS, Duman RS. A new rapid-acting antidepressant.
- 18 *Cell* **2020**;
- 19 **181(1)**:7.
- 20 29 Himmelseher S, Pfenninger E, Kochs E et al. S(+)-ketamine up-regulates neuronal
- regeneration associated proteins following glutamate injury in cultured rat hippocampal
- neurons. J Neurosurg Anesthesiol 2000;**12**:84–94.
- 23 30 Himmelseher S, Pfenninger E, Georgieff M. The effects of ketamine-isomers on
- 24 neuronal injury and regeneration in rat hippocampal neurons. Anesth Analg
- 25 1996;**83**:505–12.
- 26 31 Treccani G, Ardalan M, Chen F, et al. S-ketamine Reverses hippocampal dendritic
- Spine Deficits in Flinders Sensitive Line Rats Within 1 h of Administration. *Mol*
- 28 *Neurobiol* 2019;**56**:7368–79.
- 29 32 Höflich A, Kraus C, Pfeiffer RM, et al. Translating the immediate effects of S-ketamine
- 30 using hippocampal subfield analysis in healthy subjects-results of a randomized

- 1 controlled trial. *Transl Psychiatry* 2021;**11**:200.
- 2 33 Nummela AJ, Laaksonen LT, Laitio TT, et al. Effects of dexmedetomidine, propofol,
- 3 sevoflurane and S-ketamine on the human metabolome: A randomised trial using
- 4 nuclear magnetic resonance spectroscopy. *Eur J Anaesthesiol* 2021;**10**:1097.
- 5 34 Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, et al. Guidelines for enhanced
- 6 recovery after lung surgery: recommendations of the Enhanced Recovery After
- 7 Surgery (ERAS®) Society and the European Society of Thoracic Surgeons (ESTS).
- 8 *Eur J Cardiothorac Surg* 2019;**55**:91–115.
- 9 35 Marcantonio ER, Ngo LH, O'Connor M, et al. 3D-CAM: derivation and validation of a 3
- 10 minute diagnostic interview for CAM-defined delirium: a cross-sectional diagnostic test
- 11 study. *Ann Intern Med* 2014;**161**:554–61.
- 12 36 Mu DL, Ding PP, Zhou SZ, et al. Cross-cultural adaptation and validation
- 13 of the 3D
- 14 CAM Chinese version in surgical ICU patients. *BMC Psychiatry*
- 15 **2020;20(1)**:133.
- 16 37 Ely EW, Inouye SK, Bernard GR, et al. Delirium in mechanically ventilated patients:
- 17 validity and reliability of the confusion assessment method for the intensive care unit
- 18 (CAM-ICU). *JAMA* 2001;**286**:2703–10.
- 19 38 Inouye SK, Kosar CM, Tommet D, et al. The CAM-S: development and validation of a
- 20 new scoring system for delirium severity in 2 cohorts. Ann Intern Med 2014;160:526–
- 21 33.
- 39 Inouye SK, Leo-Summers L, Zhang Y et al. A chart-based method for identification of
- delirium: validation compared with interviewer ratings using the confusion assessment
- 24 method. *J Am Geriatr Soc* 2005;**53**:312–8.
- 40 Wang JH, Huang J, Guo FQ, et al. Circulating neurofilament light predicts cognitive
- decline in patients with post-stroke subjective cognitive impairment. Front Aging
- 27 Neurosci 2021;**13**:665981.
- 28 41 Strayer RJ, Nelson LS. Adverse events associated with ketamine for procedural
- sedation in adults. *Am J Emerg Med* 2008;**26**:985–1028.
- 42 Humeidan ML, Reyes JC, Mavarez-Martinez A, et al. Effect of cognitive prehabilitation

| 1 | on the incidence of postoperative delirium among older adults undergoing major |
|---|---|
| 2 | noncardiac surgery: the Neurobics randomized clinical trial. JAMA Surg 2021;156:148- |
| 3 | 56. |
| 4 | 43 Jung DM, Ahn HJ, Yang M, et al. Hydroxyethyl starch is associated with early |
| 5 | postoperative delirium in patients undergoing esophagectomy. J Thorac Cardiovasc |
| 6 | Surg 2018; <b>155</b> :1333–43. |
| 7 | 44 Fuchita M, Khan SH, Perkins AJ, et al. Perioperative risk factors for postoperative |
| 8 | delirium in patients undergoing esophagectomy. Ann Thorac Surg 2019;108:190–5. |
| 9 | 45 Smith PJ, Rivelli SK, Waters AM, et al. Delirium affects length of hospital stay after lung |
| 10 | transplantation. J Crit Care 2015; <b>30</b> :126–9. |
| 11 | 46 Robinson TN, Raeburn CD, Tran ZV et al. Postoperative delirium in the elderly: risk |
| 12 | factors and outcomes. Ann Surg 2009; <b>249</b> :173–8. |
| 13 | 47 Hu J, Zhu M, Gao Z, et al. Dexmedetomidine for prevention of postoperative delirium in |
| 14 | older adults undergoing oesophagectomy with total intravenous anaesthesia: A double- |
| 15 | blind, randomised clinical trial. Eur J Anaesthesiol 2021;38(Suppl 1):S9–S17. |
| 16 | 48 Perbet S, Verdonk F, Godet T, et al. Low doses of ketamine reduce delirium but not |
| 17 | opiate consumption in mechanically ventilated and sedated ICU patients: A |
| 18 | randomised double-blind control trial. Anaesth Crit Care Pain Med 2018;37:589–95. |
| 19 | 49 Kelly AM. The minimum clinically significant difference in visual analogue scale pain |
| 20 | score does not differ with severity of pain. Emerg Med J 2001;18:205-7. |
| 21 | 50 Park S, Kang CH, Hwang Y, et al. Risk factors for postoperative anxiety and depression |
| 22 | after surgical treatment for lung cancer†. Eur J Cardiothorac Surg 2016;49:e16–21. |
| 23 | 51 Wesselink EM, Kappen TH, van Klei WA, et al. Intraoperative hypotension and |
| 24 | delirium after on-pump cardiac surgery. Br J Anaesth 2015;115:427–33. |
| 25 | |
| 26 | |
| 27 | Figure legends |
| 28 | Figure 1. Consolidated Standards of Reporting Trials (CONSORT) flow |
| 29 | diagram. |

Figure 2. Overview of 3-minute Diagnostic Confusion Assessment Method

(3D-CAM) assessment.

4

5